CLINICAL TRIAL: NCT03159364
Title: Phase I/II Multicenter Trial of Antigen-specific Cytotoxic T Cells in the Treatment of Opportunistic Infections
Brief Title: Antigen-specific Cytotoxic T Cells in the Treatment of Opportunistic Infections
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17009
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Pathogen Infection; EBV Infection; CMV Infection; Adenovirus Infection; BKV Infection; Fungus Infection; Tuberculosis
Keywords: CTL; Virus CTL; Fungus CTL; TB CTL
MeSH Terms: conditions — Epstein-Barr Virus Infections; Cytomegalovirus Infections; Adenoviridae Infections; Mycoses; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infusion of pathogen-specific CTLs (Experimental): Repetitive CTL infusions to treat microbial infections
  Interventions: Biological: pathogen-specific CTLs

INTERVENTIONS:
Biological: pathogen-specific CTLs — Patients will receive approximately 1x10^5~1x10^6 CTLs/kg as a single infusion via IV injection and may receive additional infusions.

SUMMARY:
Epstein Barr Virus (EBV) or Cytomegalovirus (CMV) infection results in significant morbidity and mortality in hematopoietic stem cell transplantation (HSCT) patients. HSCT patients often face opportunistic infections due to the immunosuppressive state during transplantation. Antimicrobial drugs are usually used for prophylactic purposes and for treatment after early detectable infections. Unfortunately, some patients develop resistance to such drug treatment. In addition to HSCT patient, immune compromised patient may also be victim to opportunistic infections. Many infections can be effectively managed by functional immune recovery. In this study, the safety and efficacy of microbial-specific cytotoxic T lymphocytes (CTLs) will be investigated.

DETAILED DESCRIPTION:
Background:

Opportunistic infections are major causes of transplant-related morbidity and mortality in immunosuppressed patients, especially in the early post-transplant period. CMV, EBV, adenovirus (AdV), BK virus (BKV) and other viruses or non-viral pathogens may lead to life-threatening infections after transplantation.

Adoptive immunotherapy with cytotoxic T lymphocytes (CTLs) reactive with specific microbial antigens has proven to be effective without stimulating acute graft-versus-host disease (GVHD) owing to the significantly reduced nonspecific alloreactivity. This study aims to evaluate the safety and efficacy of treating opportunistic infections with microbial-specific CTLs in immune compromised patients.

Objective:

Primary study objectives: Infusion of autologous or allogenic pathogen-specific CTL to patients by I.V., to evaluate the safety.

Secondary study objectives: To evaluate the anti-microbial efficacy of IV-infused autologous or allogenic pathogen-specific CTLs.

Design:

Peripheral blood mononuclear cells (PBMC) will be obtained through apheresis. T cells from PBMC will be activated and enriched by dendritic cells with pathogen specific antigens. Cell preparation time is approximately 12-17 days. Subject will receive infusions of 1x105~1x106 cells/kg body weight of CTLs via IV infusion. Patients are followed weekly for one month after the infusion, monthly for 3 months, and then every 3 months until the trial ends.

ELIGIBILITY:
Inclusion Criteria:

Subjects with or without hematopoietic stem cell transplantation / organ transplant recipients need to meet the following conditions:

* Evidence of CMV, EBV, ADV, BKV or known pathogen infection (viral DNA, immunohistochemical cytology positive); contraindications or invalid to anti-microbial drugs.
* Subjects with virus DNA increased in the 2 consecutive peripheral blood samples (≥ 1000 genomic copies/ml blood) at least 24 hours apart.
* Initial hematopoietic reconstitution: neutrophils (ANC) ≥ 0.5x109 / L, platelet (PLT) ≥ 20x109 / L.
* Patients with pahogen disease (organ/ tissue infiltration) symptoms, fever, diarrhea, or lymphadenopathy, regardless of the level of peripheral blood virus DNA, and confirmed by the presence of viral DNA or microbial antigens within body fluid or biopsy.
* The subject / guardian has signed a written consent form before any trial begins.

Proper renal and hepatic functions (ULN denotes "upper limit of normal range"):

* Creatinine ≤ 2*ULN.
* Bilirubin ≤ 2*ULN.
* SGOT ≤ 3*ULN.
* SGPT≤ 3*ULN.

If CTL is not from the patient's own, then the provider of CTLs needs to meet the following criteria:

* Did not receive chemotherapy or radiotherapy within 4 weeks prior to blood collection, and did not take any steroids for the previous week, did not use Penicillin or β-lactam antibiotics, or the lowest dose of other antibiotics.
* White blood cells ≥ 3,500 / μl, lymphocytes ≥ 750 / μl.
* Obtain a signed informed consent from the patient and / or the guardian or the donor of the BMT recipient.
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or tuberculosis (TB) test is negative.
* Physical examination in line with the standard of healthy blood donors.

Exclusion Criteria:

* Subject infected with HCV (HCV antibody positive), HBV (HBsAg positive), HIV (HIV antibody positive), or HTLV (HTLV antibody positive).
* GVHD (graft-versus-host disease) performance score at II-IV.
* Subject is albumin-intolerant.
* Subject with life expectancy less than 4 weeks.
* Subject participated in other investigational somatic cell therapies within past 30 days.
* Subject with positive pregnancy test result.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Using CTCAE 4 standard to evaluate the level of adverse events after receiving autologous or allogenic pathogen-specific CTL infusion | 24 weeks
  to evaluate the level of adverse events with CTCAE 4
Viral load change after Virus-CTL infusion | 2 months
  The viral load response to the Virus-CTL infusion will be assessed by specific PCR of peripheral blood after infusion.

SECONDARY OUTCOMES:
The incidence of CTL infusion syndrome mimicking grade Ⅱ~Ⅳ GVHD within 30 days after the last dose of CTL infusion | 1 months
Reconstitution of anti-microbial immunity monitored by flow cytometry | 6 months
Number of patients with chronic GVHD-like symptom | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No